CLINICAL TRIAL: NCT05989230
Title: Emotional Awareness and Expression Therapy for People With Persistent Pain Following Orthopedic Trauma: A Pilot Feasibility Study
Brief Title: Emotional Awareness and Expression Therapy for People With Persistent Pain Following Orthopedic Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00277255; K23HD104934 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Orthopaedic Trauma; Chronic Pain; Musculoskeletal Injury
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional Awareness and Expression Therapy (Experimental): Emotional Awareness and Expression Therapy (EAET) is a non-pharmacological intervention designed to address persistent pain.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — The goal of EAET is to increase awareness of uncomfortable emotions that are often linked to stressful past experiences (e.g., anger, sadness, fear) and learn adaptive ways to experience and express those emotions, in a safe and controlled environment. Core treatment components include pain education, drawing associations between the experience of pain and emotion, and experiencing and expressing emotions via imaginary, in vivo, and real life exposures. EAET will be delivered via 8, 60-minute, weekly psychotherapy visits.
  Other Names: EAET

SUMMARY:
The purpose of this single-arm trial is to determine the feasibility of emotional awareness and expression therapy (EAET) for individuals with persistent pain following orthopedic trauma. As part of this study, participants will be asked to attend weekly EAET treatment sessions and complete assessments (including pre-treatment, post-treatment, and follow-up) consisting of questionnaires and sensory testing procedures.

DETAILED DESCRIPTION:
Orthopedic trauma, resulting in severe injuries such as multiple fractures or amputation, occurs in approximately 3 million people annually in the United States; about half of these people experience persistent pain and psychological distress (depression, anxiety, posttraumatic stress disorder [PTSD] symptoms) 6 to 12 months post injury. Pain and distress exacerbate one another, are likely to persist, and relate to disability: half of patients report substantial disability 7 years post trauma. Medical interventions such as surgery promote survival; however, there is an urgent need to develop targeted psychological interventions to treat these disabling symptoms.

Few psychological interventions are available to treat pain and distress following orthopedic trauma. Emotional Awareness and Expression Therapy (EAET) is an 8-week psychological intervention recently developed for chronic pain conditions characterized by central sensitization. EAET is unique in treating pain and mood by targeting emotion regulation processes related to traumatic life events. Such events are ubiquitous following orthopedic trauma and recent findings show that EAET results in improvements in pain and mood; thus, it may be uniquely effective to address the needs of orthopedic trauma survivors. However, there are documented barriers to implementing psychological interventions in this population, so the feasibility of EAET is unknown. The purpose of this study is to test the feasibility of delivery and assessment of EAET for orthopedic trauma survivors with persistent pain in a single-arm trial. As part of this study, participants will be asked to do the following things:

* Attend EAET treatment with a mental health provider. Session will last around 60 minutes each.
* Complete baseline, post-treatment, and follow-up assessments. These assessments will ask patients to complete questionnaires related to physical and emotional health, as well as receive sensory testing in order to examine pain processing. The questionnaires will take 20-25 minutes. The sensory testing procedures will take about 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* One or more acute orthopedic injuries
* The patient sustained an orthopedic injury including, but not limited to:

  * Pelvic or acetabulum fracture
  * Open/displaced comminuted fracture of long bones
  * Upper extremity injuries with a major nerve involvement
  * Injuries with significant injuries to major blood vessels
  * Traumatic amputation of big toe, thumb, or proximal to the wrist or ankle.
* Initial admission to the trauma or orthopedic center/service of the participating hospital OR all necessary screening and patient characteristic data available in medical record (determination based on information available at time of enrollment)
* 18 years old or older
* Received operative fixation for at least one acute orthopaedic injury at a participating hospital. Patients should be recruited at the time of primary injury, not revision or complication surgery
* Average Brief Pain Inventory Score > 3/10
* Presence of pain most days (> 3 days/week) for past three months

Exclusion Criteria:

* peri-prosthetic fractures of the femur (regardless of etiology)
* non-ambulatory due to an associated spinal cord injury
* non-ambulatory pre-injury
* currently pregnant
* moderate or severe traumatic brain injury (TBI), as evidenced by intracranial hemorrhage present on admission CT
* major amputation(s) of the upper or lower extremities
* non-English speaking
* Likely to have severe problems with maintaining follow-up for any of the following reasons:

  * The patient has been diagnosed with a severe psychiatric conditions
  * The patient has current alcohol and/or drug addiction based on medical record or patient self-report.
  * The patient is intellectually challenged without adequate family support
  * The patient lives outside the hospital's catchment area
  * The patient follow-up is planned at another medical center
  * The patient is a prisoner
  * The patient is homeless
  * Other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Enrollment | 24 months
  Feasibility of enrollment will be measured by percentage of eligible patients who enroll in the study.
Feasibility of Retention | 24 months
  Feasibility of retention will be measured by percentage of participants who are retained over the duration of the study.
Feasibility of Recruitment | 24 months
  Feasibility of Recruitment will be measured by the enrollment of a full sample within two years of the start of the enrollment period.
Percentage of patient session attendance | 8 weeks
  Percentage of patients who complete 6 of 8 total EAET sessions.
Therapist Fidelity (Questionnaire developed by study team) | 8 Weeks
  Percentage of treatment fidelity across all treatment sessions (study therapist self-report using questionnaire developed by study team).
Percentage of patients who indicate patient satisfaction and acceptability | 8 Weeks
  Percentage of patients who indicate treatment acceptability on the Treatment Evaluation Inventory-Short Form. This is a 9-item measure and participants respond using a 1-5 point likert scale for a possible total range of 9-45. Higher scores indicate greater satisfaction and acceptability.
Feasibility of Study Assessment | 1 Week
  Measured by percent of pre-treatment assessments completed by participants.
Feasibility of Study Assessment | 8 Weeks
  Measured by percent of post-treatment assessments completed by participants.
Feasibility of Study Assessment | 12 months
  Measured by percent of follow-up assessments completed by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Aaron, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ravyts SG, Carnahan N, Campbell C, Castillo R, Wegener S, Rassu FS, Lumley MA, Aaron R. Emotional awareness and expression therapy (EAET) for chronic pain following traumatic orthopaedic injury and surgery: study protocol for a single-arm feasibility clinical trial. BMJ Open. 2025 Mar 15;15(3):e093102. doi: 10.1136/bmjopen-2024-093102. PMID 40090682